CLINICAL TRIAL: NCT07222176
Title: Synergistic Effects of P-TIOX and Tixel: A Split-Face, Prospective Study
Brief Title: Effects of P-TIOX and Tixel Combined on Reducing Eye Wrinkles
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Main Line Center for Laser Surgery (Other)
Responsible Party: Principal Investigator, Kachiu Lee, MD, Principle Investigator, Main Line Center for Laser Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTIOXTIXEL
Record Dates: First submitted 2025-06-13; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Periocular Fine Wrinkles
Keywords: Periocular fine wrinkles; periocular rhytides; periocular rejuventation; tixel; skinceuticals; P-TIOX

STUDY DESIGN:
Intervention Model Description: This study utilizes a split-face, prospective, within-subject controlled design to evaluate the synergistic effects of P-TIOX combined with Tixel treatment on periocular fine lines and wrinkles.
  Each participant serves as their own control. One side of the face is randomly assigned to receive daily topical application of P-TIOX in addition to standardized Tixel treatments, while the contralateral side receives Tixel treatment alone without any topical intervention.
  This paired design allows direct comparison of treatment efficacy within the same individual, minimizing variability due to intrinsic patient factors such as skin type, lifestyle, and genetic background.
  Objective assessments using standardized imaging and blinded evaluator grading, as well as subjective patient self-assessments, are performed to evaluate differences in wrinkle severity and skin texture improvements between the two treatment sides over a 9-week study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Tixel Treatment With and Without Adjunctive P-TIOX in a Split-Face Design (Experimental): This arm involves a split-face treatment design where one side of the participant's periocular area receives a combination therapy of Tixel and topical P-TIOX, while the contralateral side receives Tixel treatment alone without any topical intervention. Tixel is a fractional thermal-mechanical device used to stimulate collagen remodeling and improve skin texture. P-TIOX is a topical cosmeceutical containing peptides and other active ingredients aimed at enhancing skin elasticity and reducing fine lines. Participants apply P-TIOX once daily to the designated side starting seven days prior to the first Tixel treatment and continuing for the duration of the 9-week study. Both sides receive standardized Tixel treatments at baseline, week 2, and week 4. The objective is to evaluate whether the addition of P-TIOX provides superior improvement in periocular fine lines and wrinkles compared to Tixel alone.
  Interventions: Combination Product: Split-Face Tixel Treatment With and Without Topical Peptide-Based Cosmeceutical (P-TIOX)

INTERVENTIONS:
Combination Product: Split-Face Tixel Treatment With and Without Topical Peptide-Based Cosmeceutical (P-TIOX) — This intervention involves applying a topical peptide-based cosmeceutical (P-TIOX) daily to one periocular area, combined with fractional thermal-mechanical treatment using the Tixel device on both sides of the face. The Tixel treatment delivers controlled heat energy to stimulate collagen remodeling and improve skin texture. One side of the face receives both P-TIOX and Tixel treatment, while the opposite side receives Tixel treatment alone, allowing comparison of the synergistic effects of the combination versus Tixel monotherapy.

SUMMARY:
This study looks at whether using a cosmeceutical called P-TIOX together with a treatment called Tixel can reduce fine lines and wrinkles around the eyes better than Tixel treatment alone. Tixel is an FDA-approved device that uses heat to improve skin texture and firmness. P-TIOX is a topical product with ingredients that may help improve the skin's appearance and elasticity.

One side of the face will be treated with both P-TIOX and Tixel, while the other side will receive Tixel only. The study will last about 9 weeks and will include several treatments and evaluations using photos and expert assessments.

Participants may notice improvement in the skin around their eyes. The results will help doctors understand if this combination treatment is more effective.

DETAILED DESCRIPTION:
This clinical trial is designed to evaluate the combined effect of a topical cosmeceutical, P-TIOX, with fractional thermal treatment using the Tixel device, on improving fine lines and wrinkles around the eyes (periocular region). The study will compare the outcomes of this combination therapy to Tixel treatment alone using a split-face design, where one side of each participant's face receives both treatments and the other side receives only Tixel.

Tixel is an FDA-cleared, fractional thermal-mechanical device that delivers controlled heat energy to the skin to stimulate collagen production and improve skin texture and elasticity. P-TIOX is an over-the-counter topical product containing a blend of peptides, acids, vitamins, and extracts that have been clinically shown to improve skin texture, elasticity, and the appearance of wrinkles.

The study will enroll 20 adult participants aged 30 years or older who have mild to moderate periocular wrinkles. Participants will be randomized to apply P-TIOX daily on one side of the face starting one week before the first Tixel treatment and continuing for the duration of the 9-week study period. Both sides will receive three standardized Tixel treatments spaced over four weeks.

Clinical outcomes will be assessed objectively by standardized photography using the Canfield Visia imaging system and analyzed by a blinded board-certified dermatologist using validated wrinkle severity scales. Subjective outcomes will be measured through patient self-assessment questionnaires. Safety will be monitored through adverse event reporting throughout the study.

This study aims to determine if combining P-TIOX with Tixel treatment provides superior improvement in periocular fine lines and wrinkles compared to Tixel alone, offering a potentially enhanced minimally invasive treatment option for facial rejuvenation.

ELIGIBILITY:
Inclusion Criteria:

* Severity of 2, 3, or 4 based on the 5-point severity scale of both periocular areas
* 30 years of age or older
* Willingness to comply with study visits
* Willingness to discontinue use of other topical cosmeceuticals/retinoids to the periocular region for the duration of the study

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior treatment with periocular laser, energy-based devices, neuromodulators, or dermal fillers within the past six months
* Prior surgical intervention in the periocular region within the past twelve months
* Use of topical retinoids in the periocular area within the past four weeks
* Known hypersensitivity to any component of P-TIOX
* Presence of active dermatologic or ocular disease in the treatment area
* Active systemic infection
* Active cold sore/herpes labialis infection

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective change in Periocular Fine Lines and Wrinkles by Canfield Visia Imaging Analysis | From baseline (Week 0) to final follow-up visit (Week 8 ± 7 days after initial Tixel treatment).
  Objective change in periocular fine lines and wrinkles will be measured using the Canfield Visia skin photography analysis system.

SECONDARY OUTCOMES:
Subjective change in Periocular Wrinkles and Texture by Dermatologist Assessment | From baseline (Week 0) to final follow-up visit (Week 8 ± 7 days after initial Tixel treatment).
  A blinded, board-certified dermatologist will evaluate pre- and post-treatment photographs using a periocular wrinkle severity scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Available upon request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available for 7 years after the conclusion of the study.
Access Criteria: Data will be available upon request.

REFERENCES:
- [Background] Bollela VR. Mind the gap! Med Educ. 2008 May;42(5):519. doi: 10.1111/j.1365-2923.2008.03073.x. No abstract available. PMID 18412894
- [Background] Sajwan RK, Solanki PR. Gold@Carbon Quantum Dots Nanocomposites Based Two-In-One Sensor: A Novel Approach for Sensitive Detection of Aminoglycosides Antibiotics in Food Samples. Food Chem. 2023 Jul 30;415:135590. doi: 10.1016/j.foodchem.2023.135590. Epub 2023 Feb 3. PMID 36870212
- [Background] Chou P, Wang GH, Hsueh SW, Yang YC, Kuo CC. Delta-Frequency Augmentation and Synchronization in Seizure Discharges and Telencephalic Transmission. iScience. 2020 Oct 9;23(11):101666. doi: 10.1016/j.isci.2020.101666. eCollection 2020 Nov 20. PMID 33134896
- [Background] Roy JM, Kazim SF, Rumalla K, Schmidt MH, Bowers CA. Geographic trends in the utilization of frailty as a preoperative decision-making tool in neurosurgery. J Neurosurg Sci. 2023 Dec;67(6):774-775. doi: 10.23736/S0390-5616.23.06104-0. Epub 2023 Jul 10. No abstract available. PMID 37428009